CLINICAL TRIAL: NCT00315029
Title: Patient-Centered Implementation of Elective Single Embryo Transfer (eSET) in in Vitro Fertilisation (IVF) and Intracytoplasmic Sperm Injection (ICSI)
Brief Title: Patient-Centered Implementation Trial for Single Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof JAM Kremer, Radboud Universty Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PITS2006; ZonMw nr 945-16-105
Record Dates: First submitted 2006-04-14; First posted 2006-04-17 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Male Infertility; Female Infertility; Pregnancy
Keywords: Implementation; Single embryo transfer; ICSI; IVF; prevention
MeSH Terms: conditions — Infertility, Male; Infertility, Female

ARMS (2):
- 1 (Experimental): Receives combined patient centred intervention
  Interventions: Behavioral: evidence based decision aid; Behavioral: Possible reimbursement 4th IVF/ICSI cycle when necessary
- 2 (No Intervention): Standard treatment

INTERVENTIONS:
Behavioral: evidence based decision aid — evidence based decision aid
  Arms: 1
Behavioral: Possible reimbursement 4th IVF/ICSI cycle when necessary — Potential reimbursement 4th IVF/ICSI cycle when necessary
  Arms: 1

SUMMARY:
Background: The number of multiple pregnancies is considered to be the most important adverse effect of in vitro fertilisation (IVF) and intracytoplasmic sperm injection (ICSI). IVF or ICSI with transferring only one embryo, elective single embryo transfer (eSET), will reduce this incidence remarkably. Unfortunately, former research has documented that cycles with SET maintain lower pregnancy rates compared to double embryo transfer (DET). Implementation of eSET will require a carefully chosen and thoroughly defined implementation strategy focussed on the couple undergoing the subfertility treatment. This trial will investigate the (cost)effectiveness of a combined patient centred implementation strategy.

Objective: The main aim is to compare the effectiveness and costs of implementation of elective single embryo transfer (eSET) in in vitro fertilisation (IVF) and intracytoplasmic sperm injection (ICSI), between usual care and a combined patient-centred strategy.

Study design: A randomised controlled trial

Study population: Couples with a female age less than 40 years ongoing an IVF/ICSI treatment in 2 of the 13 Dutch IVF centres and their 4 satellite/transport centres.

Intervention A combined patient centred implementation strategy for eSET in IVF/ICSI. The strategy consists of counselling through an evidence based decision aid and reimbursement of a 4th cycle if couples have chosen for eSET in the first 2 cycles.

Primary study parameters/outcome of the study: the eSET occurrence rate, pregnancy outcomes and cost-effectiveness of the combined strategy.

Secondary study parameters/outcome of the study:

* patient knowledge
* patient decisional conflict
* patient satisfaction
* IVF/ICSI treatment outcome.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Female age < 39 years
* In first cycle minimum of two embryos available for transfer

Exclusion Criteria:

* Medical necessity for single embryo transfer

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence choice for eSET | after embryo transfer

SECONDARY OUTCOMES:
Patient knowledge | during treatment
patient decisional conflict | during treatment
Patient experiences | duringg treatment
Pregnancy outcomes | after treatment
Cost-effectiveness | after follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rosella P Hermens, PhD, Principal Investigator — Centre for Quality of Care Research (WOK), Radboud University Nijmegen Medical Centre; Jan AM Kremer, MD, PhD, Principal Investigator — Department of Obstetrics & Gynaecology, Radboud University Nijmegen Medical Centre; Didi D Braat, Prof. MD PhD, Study Chair — Department of Obstetrics and Gynaecology, Radboud University Nijmegen Medical Centre; Richard PT Grol, Prof. PhD, Study Chair — Centre for Quality of Care Research (WOK), Radboud University Nijmegen Medical Centre; Willianne Nelen, MD, PhD, Principal Investigator — Department of Obstetrics & Gynaecology, Radboud University Nijmegen Medical Centre
Locations (2):
- Netherlands (2):
  - Catharina ziekenhuis Eindhoven, Eindhoven
  - Radboud University Nijmegen Medical Centre, Nijmegen

REFERENCES:
- [Background] Pandian Z, Templeton A, Serour G, Bhattacharya S. Number of embryos for transfer after IVF and ICSI: a Cochrane review. Hum Reprod. 2005 Oct;20(10):2681-7. doi: 10.1093/humrep/dei153. PMID 16183994
- [Background] Lukassen HG, Braat DD, Wetzels AM, Zielhuis GA, Adang EM, Scheenjes E, Kremer JA. Two cycles with single embryo transfer versus one cycle with double embryo transfer: a randomized controlled trial. Hum Reprod. 2005 Mar;20(3):702-8. doi: 10.1093/humrep/deh672. Epub 2004 Dec 23. PMID 15618254
- [Background] Lukassen HG, Schonbeck Y, Adang EM, Braat DD, Zielhuis GA, Kremer JA. Cost analysis of singleton versus twin pregnancies after in vitro fertilization. Fertil Steril. 2004 May;81(5):1240-6. doi: 10.1016/j.fertnstert.2003.10.029. PMID 15136084
- [Derived] Brabers AE, van Dijk L, Groenewegen PP, van Peperstraten AM, de Jong JD. Does a strategy to promote shared decision-making reduce medical practice variation in the choice of either single or double embryo transfer after in vitro fertilisation? A secondary analysis of a randomised controlled trial. BMJ Open. 2016 May 6;6(5):e010894. doi: 10.1136/bmjopen-2015-010894. PMID 27154481
- [Derived] van Peperstraten A, Nelen W, Grol R, Zielhuis G, Adang E, Stalmeier P, Hermens R, Kremer J. The effect of a multifaceted empowerment strategy on decision making about the number of embryos transferred in in vitro fertilisation: randomised controlled trial. BMJ. 2010 Sep 30;341:c2501. doi: 10.1136/bmj.c2501. PMID 20884700